CLINICAL TRIAL: NCT02821091
Title: Biomechanics Research in the Effects of Interactive Dynamic Balance Training on Postural and Gait Control in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limitaiotn of financial support
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201501039RINC
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2016-06

CONDITIONS: Older Adults, Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control young adults (No Intervention): Healthy adults, age between 20 to 59 yeas old
- Control old adults (No Intervention): Healthy adults, age between 60 to 80 yeas old
- Exercise old adults (Experimental): Healthy adults, age between 60 to 80 yeas old received interactive dynamic balance training
  Interventions: Other: Interactive Dynamic Balance Training

INTERVENTIONS:
Other: Interactive Dynamic Balance Training
  Arms: Exercise old adults

SUMMARY:
Aim 1: Determine the relationships between muscle quality and balance performance as well as any association with fracture and fall history in older adults.

Muscle quality will be calculated from the information of muscle strength and body composition (strength/lean muscle mass). The investigators will compute the joint torque during functional activates using biomechanical data from the 3-D motion analysis, whereas the lean skeletal muscle mass will be determined by the bioelectrical impedance analysis (BIA). Clinical and functional assessments for balance performance will also be conducted. Fracture and fall history prior to the testing will be recorded retrospectively.

Aim 2: Identify the relationships between force usages during balance perturbation in older adults.

Lateral and forward/backward perturbation while walking will be used to elicit balance recovery responses. The degree of necessary joint force and how this relates to a person's functional capacity at specific joint levels will be determined by the torque demand to capacity ratio (DCR: task demands relative to strength capacity). The DCR provides a joint-specific unified scalar quantity representing the balance recovery demand normalized by the maximum muscle strength capacity of an individual. It would indicate whether a person can recover balance and to what extent of his/her maximum capacity is taxed.

Aim 3: Examine the effectiveness and long-term effects of a novel 2-month personalized strengthening and balance training program on improving balance performance in older adults.

Personalized strengthening and balance training exercise will be personalized based on the results of biomechanical assessments, using the Modular Interactive Tiles System (MITS) and split-belt balance perturbation instrumented treadmill. The exercise group will receive training 2 times a week for 2 months and the age-matched control group will maintain their usual daily life activities. All assessments will be performed at baseline, and 1 week after training. Follow-up telephone interviews will be conducted at 6, 9, and 12 months following the training period.

DETAILED DESCRIPTION:
Aging populations has become a global issue. Fall is a prevalent concern among aging adults that can cause fracture, injury or mortality. Identifying the factors related to falls occurring within this aging population is essential for the development of effective regimes for fall prevention. Studies have shown that muscle quality and good posture alignments are critical for balance control in older adults. Older adults often combining with muscles weakness (sarcopenia), bone loss (osteoporosis) and lead to increased spine kyphosis causing vertebral fractures and poor balance control. Therefore, the long-term objectives of this work are to prevent fall in older adults by improving the function of degenerative muscles. The proposed research can provide needed information regarding the processes of balance control in this aging population, and can potentially be applied to individuals with poor balance who at high risk of fall. Three specific aims for this 3 years research project are described as follow:

Aim 1: Determine the relationships between muscle quality and balance performance as well as any association with fracture and fall history in older adults.

Muscle quality will be calculated from the information of muscle strength and body composition (strength/lean muscle mass). The investigators will compute the joint torque during functional activates using biomechanical data from the 3-D motion analysis, whereas the lean skeletal muscle mass will be determined by the bioelectrical impedance analysis (BIA). Clinical and functional assessments for balance performance will also be conducted. Fracture and fall history prior to the testing will be recorded retrospectively.

Aim 2: Identify the relationships between force usages during balance perturbation in older adults.

Lateral and forward/backward perturbation while walking will be used to elicit balance recovery responses. The degree of necessary joint force and how this relates to a person's functional capacity at specific joint levels will be determined by the torque demand to capacity ratio (DCR: task demands relative to strength capacity). The DCR provides a joint-specific unified scalar quantity representing the balance recovery demand normalized by the maximum muscle strength capacity of an individual. It would indicate whether a person can recover balance and to what extent of his/her maximum capacity is taxed.

Aim 3: Examine the effectiveness and long-term effects of a novel 2-month personalized strengthening and balance training program on improving balance performance in older adults.

Personalized strengthening and balance training exercise will be personalized based on the results of biomechanical assessments, using the Modular Interactive Tiles System (MITS) and split-belt balance perturbation instrumented treadmill. The exercise group will receive training 2 times a week for 2 months and the age-matched control group will maintain their usual daily life activities. All assessments will be performed at baseline, and 1 week after training. Follow-up telephone interviews will be conducted at 6, 9, and 12 months following the training period.

Translational research of this nature will contribute necessary information on the critical factors of balance control in older adults. The research will also test clinical innovations of exercise training to improve the long-term prognosis in this vulnerable aging population group. The unique contribution of the proposed research lies in the integration of an explicit physical examination and biomechanical approach to a relevant clinical problem within a translational model. The findings will provide a new paradigm of treatment approaches for balance control and will reduce the risk of falling and fracture. This research can potentially be applied to individuals with poor balance who are at high risk of falling.

ELIGIBILITY:
Inclusion criteria

For control young adults group:

1. able to stand and walk for 5 minutes independently without assistant
2. aging between 20 and 59 years old

For older adults group:

1. able to stand and walk for 5 minutes independently without assistant
2. aging between 60 and 80 years old;

Exclusion criteria:

1. pre-existing major lower-extremity pathology (e.g., Chronic ankle instability or severe osteoarthritis)
2. neurological disorders or balance difficulties (e.g., Vertigo, poor vision, dizziness, stroke, or epilepsy) that would prevent standing for the duration of the testing procedures without the aid of an assistive device
3. health conditions (e.g., Heart disease, uncontrolled hypertension, chronic obstructive pulmonary diseases) that would exclude participation in a balance exercise program.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2017-01-24 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan